CLINICAL TRIAL: NCT02563704
Title: A Randomized Trial of the Efficacy of Artesunate and Three Quinine Regimens in the Treatment of Severe Malaria in Children at the Ebolowa Regional Hospital - Cameroon
Brief Title: A Trial of the Efficacy of Artesunate and Three Quinine Regimens in the Treatment of Severe Malaria in Children at the Ebolowa Regional Hospital - Cameroon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, ETHE MAKA Daniel, MD, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UYaounde1
Record Dates: First submitted 2015-09-19; First posted 2015-09-30 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Malaria
Keywords: Artesunate; Quinine; Efficacy; Malaria; Children; Cameroon
MeSH Terms: conditions — Malaria | interventions — Artesunate; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ARTES (Active Comparator): * Injectable Artesunate.Each vial contained 60 mg anhydrous artesunic acid, which was dissolved in 1 ml of 5% sodium bicarbonate (provided with the drug) and then mixed with 5 ml saline solution (provided with the drug) before injecting into an indwelling intravenous catheter.
  * Patients received 2.4 mg/kg bw of parenteral artesunate at H0, H12, H24 and thereafter once daily, for a minimum of 24 hours.
  * Patients exited from the protocol if they had clinically recovered and parasitaemia was negative.
  Interventions: Drug: Artesunate
- QLD (Active Comparator): * Injectable quinine. Each vial contained 250 mg or 500 mg QB.
  * Patients received a loading dose of 16.6 mg/kg bw of QB by intravenous (IV) infusion over 4 hours followed 8 hours after the start of the loading dose, with a maintenance dose of QB at 8.3 mg/kg bw over 4 hours every 8 hours diluted in 10 ml/kg bw of 10% dextrose solution.
  * Patients received a minimum of 24 hours of parenteral treatment and exited from the protocol if they had clinically recovered and parasitaemia was negative.
  Interventions: Drug: Quinine
- QNLD3 (Active Comparator): * Injectable quinine. Each vial contained 250 mg or 500 mg QB.
  * Patients received 8.3 mg/kg bw of QB over 4 hours by IV infusion every 8 hours diluted in 10 ml/kg bw of 10% dextrose solution.
  * Patients received a minimum of 24 hours of parenteral treatment and exited from the protocol if they had clinically recovered and parasitaemia was negative.
  Interventions: Drug: Quinine
- QNLD2 (Active Comparator): * Injectable quinine. Each vial contained 250 mg or 500 mg QB.
  * Patients received 12.5 mg/kg bw of QB over 4 hours by IV infusion every 12 hours diluted in 10 ml/kg bw of 10% dextrose solution.
  * Patients received a minimum of 24 hours of parenteral treatment and exited from the protocol if they had clinically recovered and parasitaemia was negative.
  Interventions: Drug: Quinine

INTERVENTIONS:
Drug: Artesunate
  Arms: ARTES
Drug: Quinine
  Arms: QLD; QNLD2; QNLD3

SUMMARY:
The purpose of the study is to evaluate and compare the efficacy of parenteral artesunate with three quinine regimens in the treatment of severe malaria in children at the Ebolowa Regional Hospital located in the South region of Cameroon

ELIGIBILITY:
Inclusion Criteria:

* Children presenting with one or more signs of severity of malaria according to the 2013 Cameroon National Malaria Control Programme adopted criteria (impaired consciousness, abnormal behaviour, convulsions, prostration, persistent vomiting, jaundice, hyperthermia, acute respiratory distress, clinical acidosis, haemoglobinuria, cardiovascular shock, dehydration, abnormal bleeding, severe anaemia, renal impairment, hypoglycaemia and hyperparasitaemia)
* and having an initial positive parasitaemia to Plasmodium falciparum
* Other aetiologies of the presenting symptoms excluded
* Written consent from parent(s)

Exclusion Criteria:

* Prior side effects to either artesunate or quinine administration
* Severely malnourished children
* Concomitant infection

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Fever clearance time | Time (in hours) from the onset of treatment till rectal temperature went down to 37.5°C for at least 24 hour
Coma recovery time | Time (in hours) from the onset of treatment till the participant was fully conscious with a BCS of 5 or GCS of 15 for an average of 24 hours
Time to sit unsupported | Time (in hours) from the onset of treatment till when the participant could sit unsupported for an average of 24 hours if the participant was unable to do so on admission
Time to eat and drink | Time (in hours) from the onset of treatment till when the participant could eat and drink for an average of 24 hours if the participant was unable to do so on admission
Parasite clearance time | Time (in hours) from the onset of treatment to the time of the first of two successive negative blood smear through hospital discharge, an average of one week
Parasite reduction rate 24 hours after onset of treatment | 24 hours from onset of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elie MBONDA, Study Director — Faculty of Medicine and Biomedical Sciences, University of Yaounde I

REFERENCES:
- [Derived] Maka DE, Chiabi A, Obadeyi B, Mah E, Nguefack S, Nana P, Mbacham W, Mbonda E. Economic evaluation of artesunate and three quinine regimens in the treatment of severe malaria in children at the Ebolowa Regional Hospital-Cameroon: a cost analysis. Malar J. 2016 Dec 7;15(1):587. doi: 10.1186/s12936-016-1639-1. PMID 27923381